CLINICAL TRIAL: NCT07136714
Title: Is the GLP-1 Receptor Agonist Semaglutide Able to Alleviate Mood in Patients With Major Depressive Disorder and Overweight or Obesity
Brief Title: Does Semaglutide Improve Depressive Symptoms in Patients With Major Depressive Disorder and Overweight or Obesity
Acronym: SEMAMOOD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Maj Vinberg, MD, DMSc, Professor, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-511734-13-04; 2024-511734-13-04 (EU CTIS Number)
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: GLP-1; Glucagon-like peptide 1; Semaglutide; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Wegovy once--weekly s.c titrated to max dose of 2.4 mg
  Interventions: Drug: Semaglutide Injectable Product
- Placebo (Placebo Comparator): Saline s.c. once-weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Injectable Product — Semaglutide (Wegovy) once-weekly injection s.c
  Arms: Semaglutide
Drug: Placebo — Placebo (BD Posiflush) once-weekly injection s.c
  Arms: Placebo

SUMMARY:
This 26-week long, double-blinded randomized clinical trial aims to investigate the effects of semaglutide once-weekly vs. placebo on depressive symptoms in 116 patients with Major Depressive Disorder (MDD) and co-existing overweight or obesity. The treatment will be an add-on treatment to the patient's usual medication. The investigators hypothesize that adjunctive treatment with semaglutide, will lead to a significant improvement in mood compared to placebo in patients with MDD and overweight or obesity.

The primary endpoint is the change in depressive symptoms measured as difference in the 12-item self-report mood questionnaire Major Depression Inventory (MDI) from start to follow-up after 26 weeks. The MDI measures the extent to which symptoms of depression have been present in the past two weeks.

DETAILED DESCRIPTION:
This 26 week, randomized, double-blinded, placebo-controlled clinical trial investigate effects of semaglutide once-weekly vs. placebo on depressive symptoms in patients with unipolar disorder and comorbid obesity or overweight aged 18 years to 65 years. The primary endpoint is the change in depressive symptoms measured as difference in the 12-item self-report mood questionnaire Major Depression Inventory (MDI) from week 0 to week 26.

Participants will be randomized to receive once-weekly injection of either semaglutide or placebo.

Patients will be treated for 26 weeks with an initial dose of semaglutide of 0.25 mg once weekly for four weeks, 0.50 mg once weekly for four weeks 1.0 mg for four weeks, 1.7 mg for four weeks and finally 2.4 mg for the remaining treatment period. Assessments will be conducted at weeks 0, 4, 8, 12, 16, 20, 24, and 26. Adherence and adverse events will be assessed during the entire treatment period. In addition, heart rate, blood pressure, height, body weight, waist and hip circumference will be recorded. The diagnosis of depression will be confirmed at baseline and depressive symptoms will be assessed with Hamilton Depression Rating Scale (HAM-D17) at baseline week 0, 12 and 26. MDI will be completed monthly. Participants will also complete questionnaires on physical activity, cognitive complaints, perceived stress, the reward system, Quality of life, alcohol use, and sleep quality at baseline and week 26.

ELIGIBILITY:
Inclusion Criteria:

1. Informed oral and written consent.
2. Diagnosed with unipolar disorder according to the criteria of ICD10 (International Classification of Diseases, World Health Organization (WHO)) or the DSM-V (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, the American Psychiatric Association
3. Hamilton Depression Rating Scale, 17-items (HDRS-17)47 score ≥14,
4. Age 18 years to 65 years (both included)
5. Body mass index (BMI) ≥27 kg/m2
6. Able to speak and understand Danish

Exclusion Criteria:

1. Any significant medical disorder or conditions that contraindicate the investigational drug, e.g., pregnancy, presence of known allergy GLP-1 receptor agonists, severe neurological disorder, on-going drug, or alcohol abuse
2. Coercive measures
3. Females of childbearing potential who are pregnant, breast-feeding or have the intention of becoming pregnant within the next 9 months (26 weeks plus two months after discontinuation of semaglutide), or are not using contraceptives (during the whole study period) considered as highly effective (combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) intrauterine device - IUD, IUS, bilateral tubal occlusion, vasectomised partner, sexual abstinence)
4. Patients treated with corticosteroids or other hormone therapy (except oestrogens).
5. Any active substance abuse or dependence (except for nicotine)
6. Impaired hepatic function (plasma liver transaminases >2 times upper normal limit).
7. Impaired renal function (serum creatinine >150 μmol/l)
8. Cardiac problems defined as decompensated heart failure (NYHA class III/IV), unstable angina pectoris, and/or myocardial infarction within the last 12 months
9. Hypertension with systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg
10. Impaired pancreatic function (acute or chronic pancreatitis and/or plasma amylase >2 times upper normal limit). Receiving any experimental or pre-marketing drug within the last 3 months
11. Use of diabetes medication or weight-lowering pharmacotherapy e.g. semagultid within the preceding 3 months
12. Known type 1 and 2 diabetes or HbA1c>48mmol/l
13. Suicidal behaviour as judged by the investigator and based on clinical evaluation. At all contact with patient attendance (please see Table 1) possible suicidality will be evaluatedaccording to the guidelines. If the patient is evaluated as suicidal, the person will be excluded from the study and evaluated by a senior consultant in psychiatry, who will take further action.
14. Any condition that the investigator feels would interfere with trial participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | From baseline to 26 weeks of treatment
  Change in depressive symptoms measured by the Major Depression Inventory (MDI; 12-item self-report mood questionnaire). The scale ranges from 0 to 50, with higher scores indicating worse outcome.

SECONDARY OUTCOMES:
Glycaemic control parameters (blood sampling) | From baseline to 26 weeks of treatment
  Changes in HbA1c levels
Body weight | From baseline to 26 weeks
  Change in body weight in kilograms (kg).
Waist circumference | From baseline to 26 weeks of treatment
  Change in waist circumference in centimeters (cm).
Hamilton Depression Rating Scale, 17-items (HDRS-17) score | From baseline to 26 weeks of treatment
  Change in depressive symptoms measured by the Hamilton Depression Rating Scale, 17-items (HDRS-17) score. The scale ranges from 0 to 52, with higher scores indicating worse outcome.
Functioning assessment short test (FAST) score | From baseline to 26 weeks of treatment
  Changes in Functioning assessment short test (FAST) score. Total score in the range 0-72, where higher scores reflect more serious functional impairment

CONTACTS AND LOCATIONS:
Overall Officials: Maj Vinberg, MD, PhD, DMSc, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Mental Health Centre North Zealand, Hillerød, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be shared upon reasonable and relevant requests, such as for meta-analyses. All IPD will be anonymized or de-identified to protect participants' privacy and in accordance with applicable regulations, including the GDPR.
Supporting Information: Study Protocol, SAP